CLINICAL TRIAL: NCT01678521
Title: Effect of LDL-apheresis on Pentraxin3 Plasma Levels in Hypercholesterolemic Patients With Coronary Artery Disease
Brief Title: Effect of LDL-apheresis on PTX3 Plasma Levels in Hypercholesterolemic Patients
Status: Completed | Type: Observational
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Maria Grazia Zenti, principal investigator, Universita di Verona
Other Study IDs: MZentiPTX3
Record Dates: First submitted 2012-08-24; First posted 2012-09-05 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; LDL-apheresis; Coronary artery disease; PTX3; CRP; IL6; IL10
MeSH Terms: conditions — Hypercholesterolemia; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypercholesterolemic patients: Hypercholesterolemic Patients with documented CAD and poor- or non responders or intolerant to pharmacological treatment (statins) on chronic LDL-apheresis treatment
  Interventions: Procedure: LDL-apheresis

INTERVENTIONS:
Procedure: LDL-apheresis — The acronym H.E.L.P. stands for Heparin-induced Extracorporeal Low-density-lipoprotein Precipitation. Antecubital veins served as blood access. The mean blood volume processed per session is of approximately 3000 ml.
  Other Names: HELP-apheresis

SUMMARY:
Inflammation plays a major role in atherosclerosis. Pentraxin 3 (PTX3) a multifunctional pattern-recognition protein, is expressed in many tissues/cells, including innate immunity cells, endothelium and atherosclerotic plaques. Its role is controversial: it may exert protective cardiovascular effects and/or it may be an indicator of plaque vulnerability and future cardiovascular risk.

LDL-Apheresis removes apoB100-containing lipoproteins and it can prevent progression of coronary artery disease (CAD). LDL-Apheresis exerts non-lipidic beneficial effects on the procoagulatory state and on hemorheology. No data exist about the effects of LDL-Apheresis on plasma PTX3 levels.

DETAILED DESCRIPTION:
Hypercholesterolemic patients with documented CAD, on chronic fortnightly LDL-apheresis treatment will be enrolled in this study.

Blood samples will be collected before and after a single LDL-Apheresis treatment to asses PTX3, HsCRP, IL6, IL10, Fibrinogen and lipid plasma levels.

ELIGIBILITY:
Inclusion Criteria:

* Hypercholesterolemia
* documented CAD
* chronic LDL-apheresis treatment

Exclusion Criteria:

* mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypercholesterolemic patients with documented CAD, on cronic fortnightly HELP-apheresis treatment.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
acute change in PTX3 plasma values | before and at the end of one LDL-apheresis treatment (about 6 hours)
  blood samples will be collected before and after a single LDL-apheresis treatment

SECONDARY OUTCOMES:
acute change in hsCRP | before and at the end of one LDL-apheresis treatment (about 6 hours)
  blood samples will be collected before and after a single LDL-apheresis treatment
acute change in IL6 and IL10 | before and at the end of one LDL-apheresis treatment (about 6 hours)
  blood samples will be collected before and after a single LDL-apheresis treatment

CONTACTS AND LOCATIONS:
Overall Officials: Enzo Bonora, Professor, Study Director — Universita di Verona
Locations (1):
- Endocrinologia e Malattie Metaboliche, Azienda Ospedaliera Universitaria Integrata Verona, Verona, Piazzale Stefani1, Italy